CLINICAL TRIAL: NCT00967629
Title: Effect of Sevelamer Carbonate on Oxidative Stress in Patients With Diabetic Nephropathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GCO 08-0976
Record Dates: First submitted 2009-08-26; First posted 2009-08-28 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetic nephropathy; CKD progression; AGEs; oxidative stress; dietary AGEs
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Sevelamer; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevelamer Carbonate crossover (Other): Participants will be patients with stage II-IV CKD due to diabetic nephropathy randomized to start either with sevelamer carbonate or calcium carbonate
  Interventions: Drug: Sevelamer Carbonate
- Calcium Carbonate crossover (Other): Participants will be patients with stage II-IV CKD due to diabetic nephropathy randomized to start either with sevelamer carbonate or calcium carbonate
  Interventions: Drug: Calcium Carbonate

INTERVENTIONS:
Drug: Sevelamer Carbonate — This is a 4 month, prospective, comparative, crossover study. The study will be conducted in 20 patients with stage II, III or stage IV diabetic nephropathy. Patients will be randomized 1:1 to receive either 1,250 mg of calcium carbonate TID with meals (control arm) or Sevelamer Carbonate 1,600 mg (two 800 mg tablets) with meals. Each group of 10 subjects will take the assigned drug for 8 weeks. Following the 8 week treatment period, subjects will discontinue the assigned drug for a one week washout period. Following the washout period, those who were taking calcium carbonate will be crossed over to Sevelamer Carbonate therapy and those who were receiving Sevelamer Carbonate will be crossed over to calcium carbonate for a final 8 week treatment phase.
  Arms: Sevelamer Carbonate crossover
Drug: Calcium Carbonate — This is a 4 month, prospective, comparative, crossover study. The study will be conducted in 20 patients with stage II, III or stage IV diabetic nephropathy. Patients will be randomized 1:1 to receive either 1,250 mg of calcium carbonate TID with meals (control arm) or Sevelamer Carbonate 1,600 mg (two 800 mg tablets) with meals. Each group of 10 subjects will take the assigned drug for 8 weeks. Following the 8 week treatment period, subjects will discontinue the assigned drug for a one week washout period. Following the washout period, those who were taking calcium carbonate will be crossed over to Sevelamer Carbonate therapy and those who were receiving Sevelamer Carbonate will be crossed over to calcium carbonate for a final 8 week treatment phase.
  Arms: Calcium Carbonate crossover

SUMMARY:
The purpose of this study is to determine whether oral sevelamer carbonate binds advanced glycation end products (AGEs) in the gastrointestinal (GI) tract of patients with diabetic nephropathy leading to decrease body AGE load and therefore decreases the inflammation and oxidative stress in these patients.

DETAILED DESCRIPTION:
Traditional vascular risk factors alone cannot account for the elevated cardiovascular risk in patients with chronic kidney disease (CKD). In addition to a high prevalence of hypertension and diabetes, patients with CKD have elevated levels of inflammatory markers and OS, which are emerging as important risk factors for cardiovascular disease (CVD). Patients with CKD are also known to have elevated levels of circulating advanced glycation end products (AGE's), which have been shown to induce OS and to play a central role in the development of diabetic microvascular and macrovascular complications. In CKD patients, AGE's accumulate secondary to decreased renal clearance and increased endogenous production in the setting of high levels of OS. Efforts to understand relationships between the multiple vascular risk factors in chronic kidney disease may lead to reduced morbidity and mortality in this population of patients.

Sevelamer Hydrochloride is an anion exchange resin composed of multiple positively charged amine groups indicated for the treatment of hyperphosphatemia in patients with stage V CKD. The positively charged amine groups bind negatively charged dietary phosphate preventing systemic absorption. Sevelamer Hydrochloride has been shown to have the added benefits of lowering LDL levels, lowering highly sensitive C-reactive protein (hsCRP) levels, and improving insulin resistance. Patients treated with Sevelamer Hydrochloride have also been shown to have improved vascular compliance and reduced progression of coronary vascular calcification. Since AGE's are mostly negatively charged compounds, Sevelamer Carbonate by analogy, may have anti-AGE effects which could reduce inflammation and oxidative stress. Sevelamer Carbonate would have a major advantage over Calcium Carbonate-based phosphate binders, based on the fact that it would have the added advantage of reducing the levels of AGEs. The resultant reduction of both OS and inflammation would be expected to have an independent beneficial effect on the rate of progression of CKD and CVD.

We have shown in CKD patients and in animal models that AGE's correlate with levels of OS, LDL, hsCRP, and insulin resistance. Additionally, these factors can be remediated in CKD and non-CKD diabetics by decreasing overall AGE load, particularly in the diet. To date, the effect of Sevelamer Hydrochloride or Sevelamer Carbonate on OS and circulating AGE levels has not been studied. The anti-inflammatory and lipid-lowering effects of Sevelamer Hydrochloride may occur through lowering serum AGE levels and OS. Sevelamer Carbonate is an improved form of Sevelamer Hydrochloride that has been shown to be a safe and effective alternative to calcium carbonate in the treatment of hyperphosphatemia in the earlier sta'ges of CKD without causing metabolic acidosis. The development of Sevelamer Carbonate provides an opportunity to study patients with earlier stages of CKD, and to determine if it prevents or slows the progression of CKD. We propose a study designed to compare the effects of calcium carbonate and of Sevelamer Carbonate on serum AGE levels and OS in patients with stage II-IV diabetic nephropathy.

Hypothesis:

Sevelamer Carbonate administration in persons with stage II-IV CKD, compared with calcium carbonate administration, will result in at least a:

1. 20% decrease in serum levels of AGE's;
2. 10% decease in inflammatory markers of CRP and VCAM-1, or of OS (AGER1/RAGE) in circulating mononuclear cells.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Evidence of CKD II, III or IV Stage II CKD: eGFR 60-89 cc/min Stage III CKD: eGFR 30-59 cc/min Stage IV CKD: eGFR 15-20 cc/min
3. Proteinuria on urinalysis on two occasions within 18 months of recruitment
4. Diagnosis of diabetes and receiving at least one medication for diabetes mellitus.

Exclusion Criteria:

1. Age < 18 years old
2. Stage I and V CKD
3. Patients receiving active treatment for hyperphosphatemia.
4. Biopsy proven renal disease other than diabetic nephropathy
5. Hypophosphatemia
6. Hypercalcemia
7. any history of significant gastrointestinal disorders
8. any history of significant gastrointestinal surgery such as ileostomy, colostomy and colectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
serum AGE levels | baseline
  To compare the effect of Sevelamer Carbonate versus calcium carbonate on serum AGE levels in patients with stage II-IV chronic kidney disease resulting from diabetic nephropathy from baseline to 2 months and to 4 months later.
serum AGE levels | at 2 months
  To compare the effect of Sevelamer Carbonate versus calcium carbonate on serum AGE levels in patients with stage II-IV chronic kidney disease resulting from diabetic nephropathy from baseline to 2 months and to 4 months later.
serum AGE levels | at 4 months
  To compare the effect of Sevelamer Carbonate versus calcium carbonate on serum AGE levels in patients with stage II-IV chronic kidney disease resulting from diabetic nephropathy from baseline to 2 months and to 4 months later.

SECONDARY OUTCOMES:
inflammatory markers | baseline
  To compare the effect of sevelamer carbonate versus calcium carbonate on markers of inflammation, oxidative stress, and serum lipid levels in patients with stage II-IV CKD resulting from diabetic nephropathy.
inflammatory markers | at 2 months
  To compare the effect of sevelamer carbonate versus calcium carbonate on markers of inflammation, oxidative stress, and serum lipid levels in patients with stage II-IV CKD resulting from diabetic nephropathy.
inflammatory markers | at 4 months
  To compare the effect of sevelamer carbonate versus calcium carbonate on markers of inflammation, oxidative stress, and serum lipid levels in patients with stage II-IV CKD resulting from diabetic nephropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Vlassara, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Uribarri J, Peppa M, Cai W, Goldberg T, Lu M, He C, Vlassara H. Restriction of dietary glycotoxins reduces excessive advanced glycation end products in renal failure patients. J Am Soc Nephrol. 2003 Mar;14(3):728-31. doi: 10.1097/01.asn.0000051593.41395.b9. PMID 12595509
- [Background] Peppa M, Uribarri J, Cai W, Lu M, Vlassara H. Glycoxidation and inflammation in renal failure patients. Am J Kidney Dis. 2004 Apr;43(4):690-5. doi: 10.1053/j.ajkd.2003.11.022. PMID 15042546
- [Background] Goldberg T, Cai W, Peppa M, Dardaine V, Baliga BS, Uribarri J, Vlassara H. Advanced glycoxidation end products in commonly consumed foods. J Am Diet Assoc. 2004 Aug;104(8):1287-91. doi: 10.1016/j.jada.2004.05.214. PMID 15281050
- [Background] Uribarri J, Cai W, Peppa M, Goodman S, Ferrucci L, Striker G, Vlassara H. Circulating glycotoxins and dietary advanced glycation endproducts: two links to inflammatory response, oxidative stress, and aging. J Gerontol A Biol Sci Med Sci. 2007 Apr;62(4):427-33. doi: 10.1093/gerona/62.4.427. PMID 17452738